CLINICAL TRIAL: NCT02283554
Title: Platelet Rich Fibrin With 1% Metformin for the Treatment of Intrabony Defects in Chronic Periodontitis : A Randomized Controlled Clinical Trial
Brief Title: Platelet Rich Fibrin With 1% Metformin Gel for Treatment of Intrabony Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and head, department of periodontics, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014B
Record Dates: First submitted 2014-09-27; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Periodontitis
Keywords: Periodontal Surgery; Periodontal Regeneration; Growth factors; Clinical trials
MeSH Terms: conditions — Periodontitis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- ARM1- open flap debridement (OFD) (Placebo Comparator): open flap debridement done for 30 subjects. After debridement, Metformin or PRF was not added into the intrabony defect.
  Interventions: Procedure: open flap debridement (OFD)
- ARM2- open flap debridement plus PRF(Platelet rich fibrin) (Experimental): After open flap debridement, PRF( Platelet rich fibrin) was added into the intrabony defect.
  No. of subjects= 30
  Interventions: Procedure: open flap debridement (OFD); Other: Platelet rich fibrin (PRF)
- ARM3- open flap debridement plus 1%Metformin (Experimental): After open flap debridement, 1% metformin was added into the intrabony defect No. of subjects= 30
  Interventions: Procedure: open flap debridement (OFD); Drug: Metformin
- ARM4- open flap debridement plus PRF plus metformin (Experimental): After open flap debridement, PRF and 1% metformin was added into the intrabony defect.
  No. of subject- 30
  Interventions: Procedure: open flap debridement (OFD); Other: Platelet rich fibrin (PRF); Drug: Metformin

INTERVENTIONS:
Procedure: open flap debridement (OFD)
Other: Platelet rich fibrin (PRF)
  Arms: ARM2- open flap debridement plus PRF(Platelet rich fibrin); ARM4- open flap debridement plus PRF plus metformin
Drug: Metformin
  Arms: ARM3- open flap debridement plus 1%Metformin; ARM4- open flap debridement plus PRF plus metformin

SUMMARY:
ABSTRACT:

Background: Platelet-rich fibrin (PRF) is a second-generation platelet concentrate which releases various growth factors that promote tissue regeneration. Metformin (MF), a member of biguanide group has been shown to facilitate osteoblast differentiation and thus may exhibit a favourable effect on alveolar bone . Current study was designed to evaluate the combined efficacy of PRF and 1% MF gel with open flap debridement (OFD) in treatment of intrabony defects in chronic periodontitis (CP) subjects.

Methods: One hundred and twenty subjects with single defects were categorized into four treatment groups: OFD alone, OFD with PRF, OFD with 1% MF and OFD + PRF+1% MF. Clinical parameters like site specific plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), relative attachment level (RAL) and gingival marginal level (GML) were recorded at baseline before surgery and 9 months post-operatively. Percentage radiographic intra-bony defect depth reduction was evaluated using computer-aided software at baseline and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Presence of 3- wall intrabony defects ≥3 mm deep (distance between alveolar crest and base of the defect on an intraoral periapical radiograph [IOPA] ) along with an interproximal probing depth (PD) ≥5 mm after phase I therapy (scaling and root planing [SRP] ) in asymptomatic molar teeth.

Exclusion Criteria:

* Aggressive Periodontitis subjects
* Subjects with systemic conditions known to affect the periodontal status
* Medications known to affect the outcomes of periodontal therapy
* Hematological disorders and insufficient platelet count (<200,000/mm3)
* Pregnancy/lactation
* Smoking and tobacco use in any form
* Immunocompromised individuals. Those having unacceptable oral hygiene (plaque index [PI]16 > 1.5) after re-evaluation of Phase I therapy were also excluded from the study.
* In addition, teeth with furcation defects, non vital teeth, carious teeth warranting restorations and mobility of at least grade II were also excluded.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
radiographic defect depth reduction from baseline to 9 months. | radiographic defect depth reduction from baseline to 9 months.
  The primary outcome of the study was radiographic defect depth reduction from baseline to 9 months

SECONDARY OUTCOMES:
Change in PD | Assessment of PD at 3,6 and 9 months
  PD at 3,6 and 9 months was evaluated by using a UNC-15 probe from the gingival margin to the base of pockrt
Change in RAL | Assessment of RAL at 3,6 and 9 months
  RAL is measured by measuring the distance between apical level of customized acrylic stent to pocket base
Change in GML | Assessment of GML at 3,6 and 9 months
  Assessment of GML is done from apical level of customized acrylic stent, using a UNC 15 periodontal probe
Change in mSBI | Assessment of mSBI at 3,6 and 9 months
  mSBI is assessed by noting the amount of bleeding after probing, at 3,6 and 9 months
Cgange in PI | Assessment of PI at 3,6 and 9 months
  PI is assessed by noting the amount of plaque and the site of plaque present on the tooth surface at 3,6 and 9 months